CLINICAL TRIAL: NCT02568982
Title: Evolution of the Metabolic, Cardiovascular, Bone Complications and of the Quality of Life in Cushing's Disease
Brief Title: Cushing's Disease Complications
Acronym: COMPLICUSHING
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P120132
Record Dates: First submitted 2015-07-20; First posted 2015-10-06 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Cushing's Disease
Keywords: Cushing's disease; Quality of life; Metabolic; patients with Cushing's disease; cardiovascular; thromboembolic; bone complications
MeSH Terms: conditions — Pituitary ACTH Hypersecretion | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood Urinary salivary
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patient with Cushing's disease
  Interventions: Other: Exams and questionnaires

INTERVENTIONS:
Other: Exams and questionnaires — Blood sample 24hrs urinary cortisol and salivary cortisol, urinary labstick test, EKG, cardiac ultrasound, cardiac CT-scan, arterial and venous US ophthalmology examination spine X-Ray bone densitometry QoL questionnaires (SF-36, QoLCushing, Beck BDI-II)

SUMMARY:
This study aims at investigating the complications of Cushing's disease in "de novo" patients. A series of investigations will assay before treatment and every year thereafter during a 3 years follow-up period the various complications of the disease. These investigations will determine the presence and severity of cardiovascular, metabolic, and bone complications as well as the Quality of Life. Outcome of these complications after treatment, especially after pituitary surgery will be monitored, as well as cortisol levels.

DETAILED DESCRIPTION:
At inclusion the following will be investigated and recorded :

* demographic and personal medical history.
* Familial medical history related to osteoporosis, cardiovascular disorders and thromboembolism.
* Current medical treatment.
* Physical examination.
* Assessment of basal 24hrs urinary cortisol and salivary cortisol.

  - At baseline (i.e. before specific treatment of Cortisol excess):
* physical examination,
* routine biology,
* HbA1C, fasting glucose and oral glucose load,
* cholesterol, triglyceride, HDL & LDL,
* coagulation and fibrinolysis investigation,
* 24hrs urinary cortisol and salivary cortisol, urinary labstick test.
* EKG, cardiac ultrasound, cardiac CT-scan, arterial and venous US,
* ophthalmology examination,
* spine X-Ray, bone densitometry,
* QoL questionnaires (SF-36, QoLCushing, Beck BDI-II).

Every year during a 3 years follow-up the following will be investigated :

* Current medical treatment.
* Physical examination.
* Assessment of basal routine biology,
* HbA1C, fasting glucose,
* cholesterol, triglyceride, HDL & LDL,
* coagulation and fibrinolysis investigation,
* 24hrs urinary cortisol and salivary cortisol, urinary labstick test.
* EKG, cardiac ultrasound, cardiac CT-scan (if abnormal initially), arterial and venous US,
* ophthalmology examination, bone densitometry,
* QoL questionnaires (SF-36, QoLCushing, Beck BDI-II).

ELIGIBILITY:
Inclusion Criteria:

* Cushing's disease diagnosed by complementary explorations according to the National Program of Diagnosis and Care of the Cushing 's disease

Exclusion Criteria:

* other cause of Cushing's syndrome
* known inherited syndrome having for consequence an hormonal hypersecretion (NEM-1, complexe of carney, McCuneAlbright syndrome)
* patient does not understand french
* life expectancy of less than 6 months
* pregnant women
* dependent patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cushing 's disease
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
number of complications (hormonal and imaging results, quality of life) per patient (composite) | from diagnosis until 3 years of treatment
  Evaluate the frequency of :
  * metabolic complications (HbA1C, fasting glucose and oral glucose load, cholesterol, triglyceride, HDL & LDL, coagulation and fibrinolysis investigation, 24hrs urinary cortisol and salivary cortisol, urinary labstick test)
  * cardiovascular thromboembolic complications (EKG, cardiac ultrasound, cardiac CT-scan, arterial and venous US)
  * bone complications (spine X-Ray, bone densitometry)
  * quality of life alteration measured by questionnaires (SF36, QoLCushing, Beck BDI-II)

SECONDARY OUTCOMES:
Remission rate of Cushing's disease | 1 year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Bertherat, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP, Hôpital Cochin, Paris, France